CLINICAL TRIAL: NCT02409017
Title: A Comparison of Insulin Drip Protocols in Labor: A Randomized Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of time and participation in the study
Sponsor: WellSpan Health (Other)
Responsible Party: Principal Investigator, Tara L. Moore, Investigator, WellSpan Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 690224-2
Record Dates: First submitted 2015-04-02; First posted 2015-04-06 (Estimated); Last update posted 2019-10-03 (Actual); Status verified 2019-09

CONDITIONS: Diabetes; Pregnancy
Keywords: insulin drip; labor
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Protocol A (Active Comparator): Our current standard during labor
  Interventions: Procedure: Insulin drip
- Protocol B (Active Comparator): Another commonly accepted alternative for insulin drip management during labor
  Interventions: Procedure: Insulin drip

INTERVENTIONS:
Procedure: Insulin drip

SUMMARY:
To assess which of two commonly utilized insulin drip protocols has better outcomes when used during the labor process.

ELIGIBILITY:
Inclusion Criteria:

* a. Pregnant patients with either pre-existing diabetes or gestational diabetes type A2 who require insulin for euglycemia during labor and delivery

Exclusion Criteria:

* a. Those patients who decline participation
* b. Patients less than age 18 at the time of enrollment will be excluded to protect this vulnerable patient population c. Those patients who cannot be consented d. Patients scheduled for cesarean delivery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Mean maternal glucose | Labor

CONTACTS AND LOCATIONS:
Locations (1):
- WellSpan York Hospital, York, Pennsylvania, United States